CLINICAL TRIAL: NCT06861426
Title: Patients with Acute Ischemic Stroke Receiving Ginkgo Diterpene Lactone Meglumine: a Patient Registry
Brief Title: Effectiveness of Ginkgo Diterpene Lactone Meglumine in Acute Ischemic Stroke
Acronym: PIONEER
Status: Not yet recruiting | Type: Observational
Sponsor: Ying Gao (Other)
Responsible Party: Sponsor-Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Other Study IDs: 2024-DZMEC-606-01; 2022YFC3501104 (Other Grant/Funding Number: Ministry of Science and Technology of the People´s Republic of China)
Record Dates: First submitted 2025-02-27; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Ginkgo Diterpene Lactone Meglumine; Acute Ischemic Stroke; Real-World Study; Registry; Effectiveness
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GDLM group: AIS patients received GDLM and guideline-standardized treatment within 48 hours of symptom onset
  Interventions: Drug: Ginkgo Diterpene Lactone Meglumine
- Non-exposed Group: AIS patients initiated guideline-standardized treatment within 48 hours of symptom onset without exposure to Ginkgo-derived preparations.

INTERVENTIONS:
Drug: Ginkgo Diterpene Lactone Meglumine — The specific administration protocol (including time of initiation, dosage, and treatment duration) should be strictly adhered to as per the physician's prescription and meticulously documented in the case report forms (CRFs).
  Other Names: Ginkgo Diterpene Lactone Meglumine Injection; Diterpene Ginkgolides Meglumine Injection
  Groups: GDLM group

SUMMARY:
The primary purpose of this study is to investigate the effectiveness of Ginkgo Diterpene Lactone Meglumine (GDLM) for patients with acute ischemic stroke (AIS) in real-world settings.

DETAILED DESCRIPTION:
The randomized controlled trial (RCT) of GDLM for the treatment of AIS was published in JAMA Network Open, titled "Efficacy and Safety of Ginkgo Diterpene Lactone Meglumine in Acute Ischemic Stroke: A Randomized Clinical Trial." This study provided valuable insights into the efficacy and safety of GDLM in improving functional recovery for patients with AIS. However, the generalizability of these findings to real-world medical settings remains unclear, as the trial was conducted under controlled conditions that may not fully reflect routine clinical practice. To address this gap, we will conduct this study to further explore the effectiveness of GDLM in a real medical environment. Using routine clinical care data for real-world evidence, we aim to investigate the treatment's impact on a broader and more diverse patient population. This approach will allow us to better understand the practical application of GDLM in everyday clinical settings, including its potential benefits and challenges when used outside the confines of a RCT.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years, regardless of gender
* within 48 hours of stroke onset of ischemic stroke
* patient or their legally authorized representative (LAR) has signed informed consent or legally authorized oral consent with documentation

Exclusion Criteria:

* mRS score of 2 or more prior to onset
* total hospital stay less than 7 days
* use of other ginkgo-derived preparations except GDLM
* current or planned participation in any other interventional clinical trials
* inability to comply with study procedures due to documented psychiatric disorders or severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AIS patients within 48 hours of symptom onset from certified stroke centers across China
Sampling Method: Non-Probability Sample
Enrollment: 4460 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an mRS score of 0 or 1 | on day 90 after onset
  Modified Rankin Scale (mRS) is a 6-point ordinal scale from 0 [no symptoms] to 5 [severe disability] when excluding mortality, with lower scores indicating better functional outcome)

SECONDARY OUTCOMES:
Proportion of patients with an mRS score of 2 or less | on day 90 after onset
  Modified Rankin Scale (mRS) is a 6-point ordinal scale from 0 [no symptoms] to 5 [severe disability] when excluding mortality, with lower scores indicating better functional outcome)
Distribution of mRS scores | on day 90 after onset
  Modified Rankin Scale (mRS) is a 6-point ordinal scale from 0 [no symptoms] to 5 [severe disability] when excluding mortality, with lower scores indicating better functional outcome)
Incidence of new-onset stroke events (ischemic stroke or hemorrhagic stroke) | within 90 days after onset
Mortality rate | within 90 days after onset
Incidence of severe or moderate bleeding events (as defined by GUSTO criteria) | during hospital stay (up to 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, PHD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (10):
- China (10):
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Harbin Second Hospital, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jiangsu Geriatric Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Xuzhou Hospital of Traditional Chinese Medicine, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Xian Changan District Hospital, Xian, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided